CLINICAL TRIAL: NCT04778839
Title: A Phase I Study of Dose Escalation and Dose Expansion To Evaluate the Safety、Tolerability、Pharmacokinetics and Efficacy of Paclitaxel Micelles for Injection in Chinese Patients With Advanced Solid Tumor.
Brief Title: Study of Paclitaxel Micelles for Injection in Chinese Patients With Advanced Solid Tumors.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Hangzhou Dihua Biotechnology Co., LTD. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HZDH20-002
Record Dates: First submitted 2021-02-19; First posted 2021-03-03 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2024-09

CONDITIONS: Advanced Solid Tumors
Keywords: Breast cancer; ovarian cancer; non-small cell lung cancer; gastric cancer; Paclitaxel Micelles
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms | interventions — Injections; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paclitaxel Micelles for Injection (Experimental): In the First Period, Only three Participants in the first dose group were randomly assigned to 175 mg/m2 paclitaxel micelle for injection at a 1:1 rate.175 mg/m2, 260 mg/m2, 320 mg/m2, and 390 mg/m2 of paclitaxel micelle for Injection was intravenously administrated for three hours,three weeks constituted one course of treatment.
  Interventions: Drug: Paclitaxel Micelles for Injection
- Paclitaxel Injection (Active Comparator): three Participants were randomly assigned to 175 mg/m2 paclitaxel Injection,175 mg/m2 of conventional Paclitaxel Injection was intravenously administrated for three hours, three weeks constituted one course of treatment.
  Interventions: Drug: Paclitaxel injection

INTERVENTIONS:
Drug: Paclitaxel Micelles for Injection — Paclitaxel Micelles for Injection was intravenously administrated for three hours, three weeks constituted one course of treatment.
  Arms: Paclitaxel Micelles for Injection
Drug: Paclitaxel injection — Paclitaxel Injection was intravenously administrated for three hours, three weeks constituted one course of treatment.
  Arms: Paclitaxel Injection

SUMMARY:
A Phase I Study of Dose Escalation and Dose Expansion To Evaluate the Safety、Tolerability、Pharmacokinetics and Preliminary Efficacy of Paclitaxel Micelles for Injection in Chinese Patients With Advanced Solid Tumor.

DETAILED DESCRIPTION:
The study will be conducted in two parts. The first part is dose escalation and the second part is dose Expansion.During the course of dose escalation, 18-27 subjects will be enrolled to assess the safety、tolerability、pharmacokinetics、preliminary efficacy ,and determine the dose-limiting toxicity (DLT) and maximum tolerated dose(MTD) of Paclitaxel Micelles for Injection, and explore phase II clinical dosages. The second part will be adjusted according to the result of the first part. It will be divided into 4 groups, including advanced breast cancer group, ovarian cancer group, non-small cell lung cancer group and gastric cancer group, with 20 subjects in each group, to further evaluate the safety, tolerance, PK and anti-tumor activity of paclitaxel micelle.

ELIGIBILITY:
Inclusion Criteria:

* Participants are required to meet all the criteria below in order to be included in the trial:

  1. Confirmed diagnosis of advanced solid tumors by histological or cytological examination, participants have no effective standard anticancer therapy available or is failed to standard anticancer therapy.
  2. Male or female patient, aged 18 ~ 70 years.
  3. Life expectancy ≥ 3 months.
  4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
  5. Participants with at least 1 measurable tumor lesion and/or assessable non-measurable lesion based on RECIST 1.1.
  6. No radiotherapy, chemotherapy, immunotherapy or other anti-tumor therapy (such as experimental drugs, biological agents, Chinese herbal medicine, etc.), surgical treatment (except diagnostic biopsy), or complete recovery from previous surgery within 4 weeks prior to enrollment, and no surgical operation was planned during the study period.
  7. No severe hematopoietic abnormalities(no blood transfusion, no blood products, no granulocyte colony-stimulating factor, platelet stimulating factor, or other hematopoietic growth factors were corrected within 14 days prior to the screening phase laboratory examination):Hb≥90g/L , ANC≥1.5×109/L , PLT≥100×109/L.
  8. No serious organic disease of heart, liver or kidney:LVEF≥50% ; ALT(Alanine aminotransferase) or AST(Aspartate transaminase)≤2.5×upper limit of normal(ULN)(for patients with hepatic metastases, ALT or AST≤5 × ULN); TBIL(Total bilirubin)≤1.5×ULN; creatinine≤1.5×ULN and CL≥ 60 mL/min[The calculation formula was as follows: CCR (140- age)× body weight (kg) /0.818× SCR (μmol/L), and female was calculated as ×0.85].
  9. The coagulation function is normal:PT、APTT and INR≤1.5×ULN。
  10. Participants (including partners) who are willing to follow reliable contraceptive measures during the study and until 3 months after the last dosing（such as intrauterine devices [IUDs], birth control pills or condoms）.Women of child-bearing age must be negative for serum HCG within 14 days prior to study enrolment and must be non-lactating。
  11. Participants with voluntarily signature Informed Consent Form (ICF) before the test, and have a full understanding of the test content, process and possible adverse reactions.
  12. Participants with good compliance, were available for follow-up, and volunteered to comply with study regulations.

Exclusion Criteria:

* Eligible participants must not meet any of the following exclusion criteria:

  1. Patients with the toxicity of previous antitumor therapy did not return to grade 1 or below (CTCAE 5.0 grade >1, excluding toxicity such as alopecia and other toxicity judged by investigators to be of no safety risk).
  2. Patients with (including suspected) an allergic history to Paclitaxel, or any of its components, or allergic constitution (excluding mild asymptomatic seasonal allergy).
  3. Patients with bleeding tendency or who are receiving thrombolytic or anticoagulant therapy.
  4. Patients who had been treated with paclitaxel and were determined by the researchers to be resistant.
  5. Patients with active central nervous system metastases,But patients with BMs who have received prior treatment and the metastases were stable can participate in the study.
  6. Patients with cerebrovascular accident or transient ischemic attack in the previous 6 months were screened.
  7. People with active infection and need anti-infection or antiviral treatment.
  8. Patients have suffered from other malignant cancers within 5 years (except for cured basal cell carcinoma and cervical carcinoma in situ).
  9. Concomitant diseases, as determined by the investigator, that seriously endangers the safety of subjects or affects their completion of the test(such as gastrointestinal bleeding, intestinal obstruction, intestinal paralysis, interstitial pneumonia, pulmonary fibrosis, etc).
  10. Patients with a clear history of neurological or psychiatric disorders (including epilepsy and dementia).
  11. Patients who have used any drugs that is CYP2C8 and/or CYP3A4 inducer or inhibitor Within 30 days before use of the test drug(including ketoconazole and other imidazole antifungal agents, verapamil, diazepam, quinidine, cyclosporine, teniposide, etoposide, vincrine, testosterone, 17-α diethylstilbestrol, retinoic acid, quercetin, etc).
  12. Patients who received blood transfusion and transfusion of blood products, such as albumin, within 2 weeks prior to trial.
  13. Patients with peripheral neuropathy above grade II.
  14. Patients with history of myocardial infarction(within 6 months prior to enrollment) ,severe or unstable angina, coronary or peripheral artery bypass grafting or congestive heart-failure (CHF) at NYHA 3-4 level ;and patients with history of uncontrollable hypertension, arrhythmias considered clinically significant by the investigator, or electrocardiogram (ECG) abnormalities.
  15. HIV infection, or active HBV infection (HBsAg and/or HBcAb positive, with peripheral blood HBV DNA ≥1 x 103 IU/ mL), or active HCV infection (HCV antibody positive, HCV RNA≥500 IU/ mL).
  16. Alcoholics (drinking more than 14 standard units per week. 1 standard unit contains 14g alcohol,such as 360mL beer or 45mL spirits with 40% alcohol or 150mL wine)within 2 weeks before screening, or patients with drug abuse.
  17. Patients who participated in other study within the last 1 month.
  18. Pregnant or nursing women.
  19. Patients who are thought to be unsuitable for participating in the trial by the researchers because of other factors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of Paclitaxel Micelles for Injection in dose ascending and dose extension as measured by assessment of maximum tolerated dose (MTD) and dose limiting toxicity (DLT). | 2 years
  MTD was determined as the dose where more than 2 out of 6 subjects experienced DLT
The recommended dose for the phase II study | 2 years
  Determined as the recommended dose for a phase 2 study based on the adverse events and toxicities at each dose groups

SECONDARY OUTCOMES:
Cmax of Paclitaxel Micelles for Injection | Cycles 1(each cycle is 21 days) ,Day1 to Day4.
  Defined as maximum observed plasma concentration
Tmax of Paclitaxel Micelles for Injection | Cycles 1(each cycle is 21 days) ,Day1 to Day4.
  Defined as time to maximum plasma concentration
AUC0-t of Paclitaxel Micelles for Injection | Cycles 1(each cycle is 21 days), Day1 to Day4.
  Defined as area under plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration
AUC0-inf of Paclitaxel Micelles for Injection | Cycles 1(each cycle is 21 days) ,Day1 to Day4.
  Defined as area under plasma concentration-time curve from Hour 0 to infinity
λz of Paclitaxel Micelles for Injection | Cycles 1(each cycle is 21 days), Day1 to Day4.
  Defined as elimination rate constant
t½ of Paclitaxel Micelles for Injection | Cycles 1(each cycle is 21 days), Day1 to Day4.
  Defined as the apparent plasma terminal phase disposition half-life
CL of Paclitaxel Micelles for Injection | Cycles 1(each cycle is 21 days), Day1 to Day4.
  Defined as apparent clearance
Vz of Paclitaxel Micelles for Injection | Cycles 1(each cycle is 21 days), Day1 to Day4.
  Defined as apparent volume of distribution
%AUCex of Paclitaxel Micelles for Injection | Cycles 1(each cycle is 21 days), Day1 to Day4.
  Defined as AUC Extrapolated Percentage
Objective response rate (ORR) of Paclitaxel Micelles | Baseline to date of first documented progression or date of the patients drop out of the study, up to 24 months.
  PR+CR,Imaging evaluations were performed with CT/MRI chest, abdominal, and pelvic scans
Disease Control Rate (DCR) of Paclitaxel Micelles | Baseline to date of first documented progression or date of the patients drop out of the study, up to 24 months.
  PR+CR+SD,Imaging evaluations were performed with CT/MRI chest, abdominal, and pelvic scans
Progression-free survival (PFS) of Paclitaxel Micelles | Baseline to date of first documented progression or date of the patients drop out of the study, up to 24 months.
  Imaging evaluations were performed with CT/MRI chest, abdominal, and pelvic scans
Duration of remission (DOR) of Paclitaxel Micelles | Baseline to date of first documented progression or date of the patients drop out of the study, up to 24 months.
  Imaging evaluations were performed with CT/MRI chest, abdominal, and pelvic scans

CONTACTS AND LOCATIONS:
Overall Officials: jian liu, master, Principal Investigator — The First Affiliated Hospital,ZheJiang Univercity; xiaochen zhang, docter, Principal Investigator — The First Affiliated Hospital,ZheJiang Univercity
Locations (1):
- The First Affiliated Hospital,ZheJiang Univercity, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No